CLINICAL TRIAL: NCT04802694
Title: Comparison of The Effects of The Products Used In Nazogastric Tube Fixation on Skin Integrity In Babies: Randomized Controlled Study
Brief Title: The Effects of The Products Used In Nazogastric Tube Fixation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, cagri covener ozcelik, Assoc.Prof, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 87982892-929
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Skin Injury
Keywords: infant; skin; adhesives; fixation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water-based barrier tape (Experimental): The infants in experiment 1 group will be applied water-based barrier tape will be used to fix the nasogastric tube
  Interventions: Device: Water-based barrier tape
- Hydrocolloid barrier tape (Experimental): The infants in experiment 2 group, hydrocolloid barrier tape will be used to fix the nasogastric tube.
  Interventions: Device: Hydrocolloid barrier tape
- Adhesive product (Active Comparator): The silk plaster used in clinic routinely will be used for control group infants to fix the nasogastric tube.
  Interventions: Device: Silk tape

INTERVENTIONS:
Device: Water-based barrier tape — The infants in experiment 1 group will be applied water-based barrier tape. The area will be covered by water-based barrier tape to fix nasogastric tube and after waiting 1 minute for drying up it will be fastened by silk tape used in clinic. The silk tape will be 5 cm long and it will be changed in every 24 hours. Following the removal of silk tape on the water-based barrier tape, the skin integrity of the infants will be evaluated through "Neonatal Skin Condition Score Scale" and the score will be recorded in the chart. Water-based barrier tape will be applied to the area every time the plaster will be changed and current skin condition score will be noted to the chart.
  Arms: Water-based barrier tape
Device: Hydrocolloid barrier tape — As for experiment 2 group, hydrocolloid barrier tape will be used to fix the nasogastric tube. The hydrocolloid barrier tape, which was cut and shaped appropriately beforehand, will be applied to the area in order to stabilize the nasogastric tube and the tube will be stabilized with silk tape used in clinic. The silk tape will be 5 cm long and it will be changed in every 24 hours. Following the removal of silk tape on the hydrocolloid barrier tape, the skin integrity of the infants will be evaluated through "Neonatal Skin Condition Score Scale" . Since the hydrocolloid barrier tape can stay on the skin for 7 days and be transparent, the assessment of skin condition will be realized for 7 days and noted down to the chart.
  Arms: Hydrocolloid barrier tape
Device: Silk tape — The silk tape used in clinic routinely will be used for control group infants to fix the nasogastric tube without any barrier. The silk tape will be 5cm long and it will be changed in every 24 hours. Following the removal of silk tape, the skin integrity of the infants will be evaluated through "Neonatal Skin Condition Score Scale" and the score will be recorded in the chart.
  Arms: Adhesive product

SUMMARY:
The present study was planned to compare the effect of products, used in the fixation of nasogastric tube, on skin integrity of 4-6 weeks infants hospitalized at neonatal and infant units. The hypothesis of the study is "Water-based barrier tape is more effective to protect skin integrity than hydrocolloid barrier tape."

DETAILED DESCRIPTION:
The study was planned as randomized controlled and experimental design to compare the efficiency of three different methods protecting skin deficiencies using adhesive products for 4-6 weeks infants. The universe of the study consisted of 4-6 weeks infants in neonatal and infants clinics of Giresun Women's and Children's Hospital between the dates of October 2020-2021. Power analysis was performed through G*Power (v3.1.7) programme in order to determine the number of the sample. At the beginning of the study, a pilot study was carried out with 15 participants from each of the groups and the effect size was calculated as d=0.672 regarding the assessment of skin condition scores and 108 participants in total should be included in the study as 36 participants for each groups in order to obtain 80% power in the level of α=0.05. Block randomization technique is applied in the study as a randomization method. "As for data collection "Infant desciption form" and "Neonatal Skin Condition Score Scale" is used. The scale is filled by two independent observer via double-blind method.

ELIGIBILITY:
Inclusion Criteria:

* All the 4-6 weeks infants including interventional process and without any skin diseases

Exclusion Criteria:

* The infants receiving treatment without any interventional process
* Those having a skin disease
* Those infants having PICC and SVK catheters and do not meet the required criteria

Ages: 4 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-10-02 (Estimated); Study Completion 2021-10-02 (Estimated)

PRIMARY OUTCOMES:
Water-based barrier tape | 24 hours
  To evaluate the skin integrity of the infants following the removal of silk adhesive from water-based barrier tape
Hydrocolloid barrier tape | 24 hours
  To evaluate the skin integrity of the infants following the removal of silk adhesive from hydrocolloid barrier tape
Adhesive tape | 24 hours
  To evaluate the skin integrity of the infants following the removal of silk adhesive from infants skin without any barrier tape

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun University Women and Children's Hospital, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lund CH, Osborne JW. Validity and reliability of the neonatal skin condition score. J Obstet Gynecol Neonatal Nurs. 2004 May-Jun;33(3):320-7. doi: 10.1177/0884217504265174. PMID 15180195